CLINICAL TRIAL: NCT00753532
Title: A Double Blind Placebo Controlled Study On The Neuroprotective And Anti-Atherogenic Effects Of Palm TocotrienolRich Fraction(Palm Vitamin E)
Brief Title: Neuroprotective and Cardioprotective Effects Of Palm Vitamin E Tocotrienols
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Malaysia Palm Oil Board (Other Government)
Responsible Party: Principal Investigator, Yuen Kah Hay, Professor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MPOB-USM-Version 1.4
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Cerebrovascular Disorders
Keywords: Carotid artery stenoses; Brain ischaemia; stroke; Lipid abnormalities; Fatty Liver
MeSH Terms: conditions — Cerebrovascular Disorders; Carotid Stenosis; Stroke; Fatty Liver | interventions — Tocotrienols; Tocovid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI(+ve), (Placebo Comparator): 121 volunteers in MRI(+ve) cohort were randomized into two groups to receive either 200mg palm vitamin E (tocotrienols) softgel capsules or a identical looking placebo twice daily. 62 volunteers received 200mg palm vitamin E (tocotrienols) and the remaining 59 received placebo. They were followed up every 3 months for a period of 2 years for their blood biochemistry profile and MRI of the brain was conducted at baseline, 12 months and 24 months..
  Interventions: Dietary Supplement: 200mg of Palm vitamin E (tocotrienols) or placebo
- MRI(-ve) (Placebo Comparator): 120 volunteers in MRI(-ve) cohort were randomized into two groups to receive either 200mg palm vitamin E (tocotrienols) softgel capsules or a identical looking placebo twice daily. 63 volunteers received 200mg palm vitamin E (tocotrienols) and the remaining 57 received placebo. They were followed up every 3 months for a period of 1 year for their blood biochemistry profile and MRI of the brain was conducted at baseline and 12 months.
  Interventions: Dietary Supplement: 200mg of Palm vitamin E (tocotrienols) or placebo

INTERVENTIONS:
Dietary Supplement: 200mg of Palm vitamin E (tocotrienols) or placebo — Individuals randomized in the (MRI+ve) and (MRI -ve) cohort respectively. In the MRI(+ve) cohort, 62 subjects received 200 mg softgels of Palm Vitamin E (tocotrienols) and 59 were assigned to placebo, taken orally twice a day for a study period of two years. In the MRI(-ve) cohort, 63 subjects received 200 mg softgels of Palm Vitamin E (tocotrienols) and 57 consumed placebo, taken twice a day for a follow up period of 1 year.
  Other Names: Tocovid 200mg

SUMMARY:
The purpose of the study is to assess the neuroprotective, anti atherogenic and hepatoprotective properties of tocotrienols (palm vitamin E) supplementation as determined by white matter lesion load on serial magnetic resonance imaging (MRI), carotid artery magnetic resonance angiography (MRA) and liver ultrasound (US) as well as lipid profile analysis.

DETAILED DESCRIPTION:
Stroke is the third largest cause of death after heart disease and cancer in Malaysia. It is estimated that 52,000 Malaysians suffer stroke annually. In 2005, 3245 cases of stroke were fatal. It is projected that the number of fatal stoke cases will exceed 25,000 in 2020.

It was found that at nanomolar concentrations, α-tocotrienol but not α-tocopherol prevent glutamate-induced neuron cell death in mice through inhibition of c-Src kinase and 12-lipoxygenase. Tocotrienol-supplemented rats showed more protection against stroke-induced injury compared with matched controls.

White matter lesion as detected on magnetic resonance imaging (MRI) is closely related to vascular events of the brain. MRI and histopathological study has shown that the larger white matter lesions not usually conforming to usual areas infarcts can actually represent areas of subclinical infarct. In addition there is positive correlation between white matter lesions with established vascular risk factors.

The Rotterdam Scan Study showed that elderly people with silent brain infarcts and white matter lesions are at a strongly increased risk of clinical stroke, which could not be explained by the major stroke risk factors alone.

Several recent studies showed that white matter lesions may be an independent prognostic measure of future stroke risk.

White matter hyperintensities as detected on MRI is closely related to vascular events of the brain and in some instances represent subclinical infarcts.

It is therefore conceivable to study the neuroprotective properties of tocotrienol supplementation in humans by looking at serial changes of white matter disease load.

Tocotrienol supplementation brings about various favourable effects including improving lipid profiles, lowering of thromboxane B2 and platelet factor 4 and reduced LDL oxidation. Carotid artery MR angiography is an established and robust technique in the evaluation of carotid artery stenosis. Therefore, to study the anti-atherogenic effects of tocotrienols supplementation, serial MR angiography of the carotid arteries are done.

Non-alcoholic fatty liver disease (NAFLD) is emerging as a not fully understood, both in aetiology and significance, liver disorder. FLD is reported to be the most common cause of chronic liver disease in the U.S.A. and other western countries with a prevalence rate ranging between 15% to 30% of the adult population. However, limited data are available for Malaysia.

US imaging provides valuable information of the liver condition with a sensitivity of 93-100%. Frequently NAFLD is associated with dyslipidemia, obesity, insulin resistance and type II diabetes and it represents the liver component of the metabolic syndrome (MetS). Patients with NAFLD are reported to have low levels of serum vitamin E. NAFLD patients present a significant increase in cardiovascular (CV) risk, thus linking NAFLD, MetS and accelerated atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Participant able to understand and has signed and dated the Informed Consent Form
* Participant can be either a male or female
* Participant is more than 35 years of age
* Participant has total cholesterol between 5.2 - 6.2 mmol/L and LDL cholesterol between 2.6 - 4.2 mmol/L
* Participant is able to comply with visits and medications
* Participant has normal liver function (total protein, total albumin, total globulin, total bilirubin, SGOT and SGPT)

Participants who satisfy the Inclusion and Exclusion Criteria for Study in General with one or more of the following conditions will be eligible for MRI screening:

* More than 40 years of age
* Stable hypertension requiring only out-patient management
* Diabetes mellitus requiring only out-patient management
* Ischaemic heart disease requiring only out-patient management
* Body mass index more than 25 (overweight or obese)

Exclusion Criteria:

* Female participants who are pregnant
* Participant has previously received vitamin E supplementation (tocotrienols or tocopherols) within the past 3 months at the time of recruitment
* Participant has a history of cancer or has undergone radiation therapy
* Participant has a history of major organ dysfunction, such as moderate or severe hepatic impairment, severe renal insufficiency, severe or unstable cardiovascular, respiratory, hematological, endocrinological, neurological or other somatic disorders resulting in previous hospitalization.
* Participant has a neurological impairment or psychiatric disorder preventing his understanding of consent and his ability to comply with the protocol.
* Participant is requiring long term anti-epileptics, hypnotics, and chronic medications for hypercholesterolemia
* Participant has very high cholesterol levels, total cholesterol above 6.2 mmol/L and LDL cholesterol above 4.2 mmol/L, which require medical treatment.
* Participant is requiring long term non-steroidal anti-inflammatory (NSAID) medication.
* Participant has a history of hypersensitivity to vitamin E.
* Participant has signs of alcohol and drug dependence or abuse.
* Participant is unable to understand and comply with the elements in the consent form.

In addition, the participant must not have any contraindication to have MRI examinations including:

* Biostimulators (e.g. cardiac pacemaker and implanted spinal cord stimulator)
* Neurostimulators
* Aneurysm clips in the brain
* Cochlear implants
* Hearing aids
* Orthopaedic implants less than 2 months old
* Metal fragments in eyes Any further implants or foreign body not listed above should have the safety assessed by a radiologist prior to recruitment into the MRI study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2007-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Regression of white matter lesion load in terms of numbers and size in the brain | 1 to 2 years

SECONDARY OUTCOMES:
Regression of the carotid artery stenoses in terms of percentage | 1 to 2 years
The improvement in the lipid profile other markers associated with increased cardiovascular risk | 1 to 2 years
Improvement in liver echogenicity. | 1 to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuen Kah Hay, Phd, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Kepala Batas Hospital, Kepala Batas, Pulau Pinang, Malaysia

REFERENCES:
- [Derived] Gopalan Y, Shuaib IL, Magosso E, Ansari MA, Abu Bakar MR, Wong JW, Khan NA, Liong WC, Sundram K, Ng BH, Karuthan C, Yuen KH. Clinical investigation of the protective effects of palm vitamin E tocotrienols on brain white matter. Stroke. 2014 May;45(5):1422-8. doi: 10.1161/STROKEAHA.113.004449. Epub 2014 Apr 3. PMID 24699052
- [Derived] Magosso E, Ansari MA, Gopalan Y, Shuaib IL, Wong JW, Khan NA, Abu Bakar MR, Ng BH, Yuen KH. Tocotrienols for normalisation of hepatic echogenic response in nonalcoholic fatty liver: a randomised placebo-controlled clinical trial. Nutr J. 2013 Dec 27;12(1):166. doi: 10.1186/1475-2891-12-166. PMID 24373555